CLINICAL TRIAL: NCT02091388
Title: A Randomized, Open-Label, Parallel-Group Study to Assess the Relative Bioavailability of LY03004 and Risperdal® Consta® at 25 mg Following Multiple Intramuscular Injections in Stable Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Bioavailability of LY03004 and Risperdal® Consta®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY03004 MD
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY03004 25 mg (Experimental): 5 intramuscular injections 25 mg over 113 days
  Interventions: Drug: LY03004
- Risperdal® Consta® 25 mg (Active Comparator): 5 intramuscular injections 25 mg over 113 days
  Interventions: Drug: Risperdal® Consta®

INTERVENTIONS:
Drug: LY03004
  Arms: LY03004 25 mg
Drug: Risperdal® Consta®
  Arms: Risperdal® Consta® 25 mg

SUMMARY:
This study is to assess the bioavailability of LY03004 compared to Risperdal Consta as well as the evaluate the safety and tolerability and preliminary efficacy of LY03004 with repeat injections

DETAILED DESCRIPTION:
* To assess the relative bioavailability of LY03004 compared to Risperdal® Consta® at 25 mg following multiple intramuscular injections at steady-state;
* To evaluate the safety and tolerability of LY03004 following repeated intramuscular injections
* To evaluate the preliminary efficacy of LY03004 following repeated intramuscular injections

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 65 years old
2. Patients must have a DSM-IV-TR diagnosis of schizophrenia or schizoaffective disorder based on the Mini-International Neuropsychiatric Interview (MINI)
3. Patients must be clinically stable on antipsychotic medications other than risperidone or paliperidone or clozapine for at least 4 weeks prior to screening, based on clinical assessments AND a Positive and Negative Syndrome Scale (PANSS) total score less than or equal 70 at Screening Visit
4. Patients with a Body Mass Index in range of 18.0 to 35.0
5. Patients with an Informed Consent Form signed by the patient or legally authorized representative

Exclusion Criteria:

1. Patients with a mental disorders other than schizophrenia or schizoaffective disorder, according to the DSM-IV-TR
2. Patients who received oral risperidone or paliperidone or clozapine within 14 days prior to screening, or Risperdal® Consta® within 100 days prior to screening or paliperidone palmitate within 10 months prior to screening
3. Patients with neuroleptic malignant syndrome or physical fatigue associated with dehydration or malnutrition
4. Patients who pose a significant risk of a suicide attempt based on history, investigator's judgment or have answered "yes" to the questions 4 or 5 for current or past 30 days on the screening form of the Columbia Suicide Severity Rating Scale (C-SSRS)
5. Patients with a history of sensitivity to akathisia and other EPS, especially with previous use of risperidone or paliperidone
6. Patients with uncontrolled diabetes mellitus as indicated by a HbA1c level greater than or equal to 7%
7. Patients with a history of or currently having epilepsy or convulsion disorders
8. Patients who have had electroconvulsive therapy within the past 2 months prior to screening
9. Patients who used medication known to be an inducer or inhibitor for CYP 2D6 within 2 weeks prior to screening
10. Patients with a history of allergic reaction to risperidone or to the excipients of LY03004
11. Patients who have met DSM-IV-TR criteria for substance abuse or dependence with the exception of caffeine or nicotine in the past 6 months prior to screening
12. Patients with a history of clinically relevant cardiac arrhythmia's, cardiovascular disease, thyrotoxicosis, parkinsonism, or hemorrhagic diathesis
13. Patients who are currently taking medications with primarily CNS activities such as antidepressants, mood stabilizers or anticonvulsants
14. Patients who have participated in a clinical trial of another investigational drug within 30 days prior to screening
15. Female patients who are pregnant or are breastfeeding or are of childbearing potential without adequate use of contraception
16. Patients who have any clinically relevant hepatic, renal and cardiac dysfunction, or other medical condition or laboratory abnormality, which in the judgment of the investigator would interfere with the subject's ability to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cmax, Tmax, for Relative bioavailability of LY03004 compared to Risperdal® Consta® | 113 Days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 113 Days
The change of the PANSS score for the Preliminary efficacy of LY03004 | 113 Days

CONTACTS AND LOCATIONS:
Overall Officials: Simon Li, Study Chair — Luye Pharma Group Ltd.
Locations (10):
- United States (10):
  - Woodland International, Little Rock, Arkansas
  - Collaborative Neuroscience Network LLC, Long Beach, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - Comprehensive Clinical Development, Washington D.C., District of Columbia
  - Compass Research, Leesburg, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CBH Health LLC, Rockville, Maryland
  - CRI LifeTree, Marlton, New Jersey
  - CRI LifeTree, Philadelphia, Pennsylvania
  - Community Clinical Research Inc, Austin, Texas

REFERENCES:
- [Derived] Wang W, Wang X, Dong Y, Walling DP, Liu P, Liu W, Shi Y, Sun K. Population Pharmacokinetic Analysis to Support and Facilitate Switching from Risperidone Formulations to Rykindo in Patients with Schizophrenia. Neurol Ther. 2024 Apr;13(2):355-372. doi: 10.1007/s40120-024-00578-w. Epub 2024 Jan 20. PMID 38244179